CLINICAL TRIAL: NCT04050579
Title: A Single Center Trial of On-pump Intracardiac Echocardiography (OPIE) in the Thin Interventricular Septum
Brief Title: OPIE in the Thin Interventricular Septum
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was determined to be focused on Quality Assurance (QA) and Quality Improvement (QI), rather than research, based on its primary purpose and activities. Study was closed prior to enrollment.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: s19-01180
Record Dates: First submitted 2019-08-06; First posted 2019-08-08 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Hypertrophic Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- OPIE in thin inverventricular septum (Other): The Principal Investigator use the OPIE probe to measure the anterior basilar septal thickness. Myectomy will be performed and OPIE will be repeated.
  Interventions: Device: on-pump intracardiac echocardiography

INTERVENTIONS:
Device: on-pump intracardiac echocardiography — Subjects will be patients with hypertrophic cardiomyopathy with interventricular septae less than 2.0cm who are undergoing septal myectomy. The patients will have already had a number of preoperative transthoracic echocardiographs as part of their normal hypertrophic cardiomyopathy care. Before cardiopulmonary bypass, the basal anterior septal thickness will be measured by transesophageal echocardiograph as is performed in all septal myectomy procedures. The Principal Investigator will then use the OPIE probe to measure the anterior basilar septal thickness. Myectomy will be performed and OPIE will be repeated. The post-myectomy anterior basilar septal thickness will again be measured by transesophageal echocardiography.

SUMMARY:
This is a follow up investigation to our previous study entitled "On-pump intraoperative echocardiography (OPIE)" (clinicaltrials.gov NCT03094325) whereby we determined that left ventricular septal thickness as measured by the OPIE technique correlates highly with traditional methods of transthoracic and transesophageal echocardiography during septal myectomy for hypertrophic cardiomyopathy. OPIE may be especially useful in patients with a thin ventricular septal thickness as adequate treatment may rely on mere millimeters of myocardial resection. We therefore propose a study in which OPIE is compared to transthoracic and transesophageal echocardiography in patients with a thin interventricular septum. Subjects will receive the same perioperative care regardless of their involvement in the study. Patients who enroll in the study will undergo an additional intraoperative echocardiographic measurement that adds less than five minutes to total operative time.

ELIGIBILITY:
Inclusion Criteria:

* All hypertrophic cardiomyopathy patients, inclusive of male and female and all racial/ethnic origins, age 18 or older who are scheduled to receive a septal myectomy with a preoperative transthoracic echocardiograph suggesting an interventricular septal width of less than 2.0 cm.

Exclusion Criteria:

* Those hypertrophic cardiomyopathy patients who are scheduled to receive a septal myectomy who are less than 18 years old or whose preoperative transthoracic echocardiograph suggests an interventricular septal width of greater than 2.0 cm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2025-05-20 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
correlations | at the conclusion of all data collection; approximately 6 to 12 months
  correlation between OPIE and traditional imaging methods

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Swistel, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with New York University Langone Health. Requests may be directed to: daniel.swistel@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.

REFERENCES:
- [Background] Williams DM, Nampi RG, Saric M, Grossi EA, Sherrid MV, Swistel DG. A novel imaging modality to guide septal myectomy for hypertrophic cardiomyopathy. Podium presentation at the Western Thoracic Surgical Society Association Annual Meeting. Squaw Valley, CA. June 28, 2019.